CLINICAL TRIAL: NCT00825487
Title: A Phase 1 Dose Escalation Study of ARQ 621 in Adult Patients With Metastatic Solid Tumors and Hematologic Malignancies
Brief Title: Dose Escalation Study of ARQ 621 in Adult Patients With Metastatic Solid Tumors and Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 621-101
Record Dates: First submitted 2009-01-13; First posted 2009-01-21 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Metastatic Solid Tumors, Refractory/Relapsed Hematologic Malignancies
Keywords: metastatic; hematologic; malignancy; multiple; myeloma; malignant; lymphoma; chronic; lymphocytic; leukemia; acute; myelogenous; promyelocytic; dose escalation; safety; tolerability; pharmacodynamics; tumor; PK
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasm Metastasis; Neoplasms; Neoplasms, Plasma Cell; Lymphoma; Bronchiolitis Obliterans Syndrome; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 621 treatment (Experimental)
  Interventions: Drug: ARQ 621

INTERVENTIONS:
Drug: ARQ 621 — Treatment will be initiated at a dose level of 10 mg/m^2 IV infusion for an hour once weekly in 4-week (28 day) consecutive and continuous cycles. ARQ 621 should be infused IV over two hours at doses 200 mg/m^2 and higher (cohort 8 and above).

SUMMARY:
This is an open-label, dose escalation study of intravenous ARQ 621 administered to patients with late-stage solid tumors or hematologic malignancies.

DETAILED DESCRIPTION:
The study is designed to explore the safety, tolerability and pharmacokinetics of ARQ 621 and define a recommended phase 2 (RP2D)dose of ARQ 621.Treatment will be initiated at a dose level of 10 mg/m^2 IV infusion for an hour once weekly in 4-week (28 day) consecutive and continuous cycles. ARQ 621 should be infused IV over two hours at doses 200 mg/m^2 and higher (cohort 8 and above). All cycles of therapy will consist of the patient taking ARQ 621 intravenously once weekly for 4 weeks. Dose escalation will proceed initially by doubling (cohorts 2 and 3) and subsequently by a modified Fibonacci scheme. Dose escalations will be performed using 3-6 patient cohorts. In these cohorts, if a single dose limiting toxicity (DLT) is experienced among patients 1-3, the dose cohort will be expanded to six patients. The maximum tolerated dose (MTD) will be defined as the dose level at which no greater than 1/6 patients experiences a DLT. Once an MTD is identified, up to an additional 20 patients (with types of malignancy to be determined at a later date by study investigator and clarified by study amendment) may be treated at this MTD of ARQ 621. If an MTD is not identified in the initial 10 dosing cohorts, dose escalation will proceed in a manner to be defined by subsequent amendment with the purpose of determining a RP2D of ARQ 621.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained and documented according to International Conference on Harmonisation (ICH)- Good Clinical Practice (GCP), the local regulatory requirements, and permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPPA) prior to study-specific screening procedures
* A histologically or cytologically confirmed metastatic solid tumor or refractory/relapsed hematologic malignancy
* Have a life expectancy of at least 12 weeks
* ≥18 years of age
* Measurable disease as defined by:

  * Solid Tumors: Response Evaluation Criteria in Solid Tumors
  * Multiple Myeloma (MM): International Uniform Response Criteria, at least one of the following:

    * Monoclonal protein in the plasma of ≥0.5 g/dL
    * Monoclonal protein in the urine of ≥0.2 g/24 hr urine collection
    * Serum immunoglobulin free light chain (FLC) ≥100 mg/L (10 mg/dL) and abnormal serum immunoglobulin kappa to lambda FLC ratio
  * Malignant Lymphoma (ML): International Working Group Response Criteria

    * At least one site of disease ≥2 cm in longest diameter (a lesion ≥1 cm can be considered if PET positive)
  * Chronic Lymphocytic Leukemia (CLL): NCI Working Group Guidelines

    * Lymphocytosis (5 x 10^9 /L) with B-cell marker (CD19, CD20,CD23) + CD5
    * High-risk characteristics (hemoglobin <10g/dL OR platelets <100 x 10^9 /L)
  * Acute Myelogenous Leukemia (AML) or Acute Lymphoblastic Leukemia (ALL): only patients with bone marrow or peripheral blast count of ≥20%
  * Acute Promyelocytic Leukemia (APML): patients must be refractory to all-trans retinoic acid (ATRA) and arsenic trioxide
  * Chronic Myelogenous Leukemia (CML): patients in blast crisis (bone marrow or peripheral blast count ≥20%) may be included if refractory to prior therapy and to any therapy the investigators deems of higher priority (for example, BCR-ABL inhibitors such as imatinib mesylate [Gleevec], nilotinib [Tasigna], or dasatinib [Sprycel])
* ECOG performance status ≤2
* Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last ARQ 621 dose
* Females of childbearing potential must have a negative serum pregnancy test
* Aspartate transaminase (AST) and alanine transaminase (ALT) ≤2.5 × upper limit of normal (ULN) or ≤5.0 × ULN with metastatic liver disease
* Hemoglobin (Hgb) ≥10 g/dL (except in cases considered related to hematologic malignancy)
* Total bilirubin ≤1.5 × ULN
* Creatinine ≤1.5 x ULN (≤2.0 x ULN in cases considered related to multiple myeloma)
* Absolute neutrophil count ≥1.5 x 10^9/L (except in cases considered related to hematologic malignancy)
* Platelets ≥100 x 10^9/L (except in cases considered related to hematologic malignancy)
* Patients with hematologic malignancies who have progressed following at least two prior treatment regimens

Exclusion Criteria:

* Anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents within four weeks of the first dose

  * In cases of hematologic malignancies, 4-week recovery from prior anticancer treatment is not required, however the patient must recover from prior treatment-related non-hematological toxicities to grade 2 or less
  * When required for supportive care corticosteroids or hydroxyurea may be used
* Surgery within four weeks prior to the first dose
* Known untreated brain metastases or leptomeningeal disease

  * Patients with solid tumors who were treated for brain metastases and who have shown stable disease for at least 8 weeks prior to enrollment will be allowed
* Pregnant or breastfeeding
* Uncontrolled concurrent illness including, but not limited to ongoing or active symptomatic infection requiring systemic therapy, clinically significant non-healing or healing wounds, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements
* Patients having a history of Thrombotic thrombocytopenic purpura (TTP) or Hemolytic-uremic syndrome (HUS) or HUS spectrum will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the safety, tolerability and recommended Phase 2 dose (RP2D) of ARQ 621 administered intravenously. | 24 months estimated

SECONDARY OUTCOMES:
To determine the pharmacokinetic profile of ARQ 621. | 24 months estimated
To determine the pharmacodynamic profile (incl. biomarkers) of ARQ 621. | 24 months estimated
To assess the preliminary anti-tumor activity of ARQ 621. | 24 months estimated

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Translational Genomics Institute, Phoenix, Arizona
  - Premiere Oncology, Santa Monica, California
  - Boston, Massachusetts
  - Nevada Cancer Institute, Las Vegas, Nevada